CLINICAL TRIAL: NCT05034185
Title: Real-World Validation of an Artificial Intelligence Characterization Support (CADx) System for Prediction of Polyp Histology in Colonoscopy: A Prospective Multicentre Study
Brief Title: Real-World Validation of an Artificial Intelligence Characterization Support (CADx) System
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore General Hospital (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, James Li Weiquan, Consultant, Changi General Hospital
Other Study IDs: CIRB Ref: 2021/2001
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Dysplasia
Keywords: colonoscopy; computer-aided diagnosis; colorectal polyp; colorectal neoplasm; artificial intelligence
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms; Colorectal Neoplasms | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colorectal polyps detected during colonoscopy will be resected for final histology, which will form the gold standard for evaluation of the diagnostic accuracy of the Clinician using IEE versus the CADx support tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with one or more polyps detected: During colonoscopy, the Clinician inspect for the presence of polyps as per routine clinical practice with the CAD EYE function turned off. When a polyp is encountered, the Clinician will make a prediction on the histology based on the white light and BLI features of the polyp with and without optical magnification, as per routine clinical practice. Following this, the CAD EYE function will be switched on and the Clinician will take note of the CADx prediction for the same polyp, which will be either "neoplastic" or "hyperplastic".
  In addition, other polyp features such as the size and location will be recorded, which is similar to what is performed in routine clinical practice. The polyp will be resected and sent for pathological examination, which will form the "gold standard" for the diagnosis of polyp histology.
  Interventions: Device: Computer-aided diagnosis (CADx) support tool

INTERVENTIONS:
Device: Computer-aided diagnosis (CADx) support tool — The CADx support tool operates when the Clinician switches the preconfigured CAD EYE function on using a button on the controller while the scope system is in BLI mode. This is performed after the Clinician first makes an optical prediction of polyp histology using IEE as described. The CADx support tool will make a prediction of polyp histology as "hyperplastic" or "neoplastic".

SUMMARY:
Colorectal cancer (CRC) is a leading cause of cancer-related morbidity and mortality worldwide, with rates of CRC predicted to increase. Colonoscopy is currently the gold standard of screening for CRC. Artificial intelligence (AI) is seen as a solution to bridge this gap in adenoma detection, which is a quality indicator in colonoscopy. AI systems utilize deep neural networks to enable computer-aided detection (CADe) and computer-aided classification (CADx). CADe is concerned with the detection of polyps during colonoscopy, which in turn is postulated to help decrease the adenoma miss-rate.

In contrast, CADx deals with the interpretation of polyp appearance during colonoscopy to determine the predicted histology. Prediction of polyp histology is crucial in helping Clinicians decide on a "resect and discard" or "diagnose and leave strategy". It is also useful for the Clinician to be aware of the predicted histology of a colorectal polyp in determining the appropriate method of resection in terms of safety and efficacy. While CADe has been studied extensively in randomized controlled trials, there is a lack of prospective data validating the use of CADx in a clinical setting to predict polyp histology.

The investigators plan to conduct a prospective, multi-centre clinical trial to validate the accuracy of CADx support for prediction of polyp histology in real-time colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is currently the gold standard of screening for CRC. A 1% increase in adenoma detection rate (ADR) estimated to be associated with a 3% decreased risk of interval CRC. AI systems can be broadly divided into CADe (for detection) and CADx (for diagnosis, or prediction of polyp histology in the context of colonoscopy). CADe has been extensively studied, with several randomized controlled trials and meta-analysis showing a higher ADR when CADe is used compared to the control groups without CADe.

Besides the ADR, predicted polyp histology is a key component in the performance of colonoscopy as this enables the Clinician to make a decision regarding its management, as described above. In this regards, image-enhanced endoscopy (IEE) is often used to help Clinicians determine if colorectal polyps found on colonoscopy are neoplastic or hyperplastic. The most commonly used non-magnification classification is the NBI International Colorectal Endoscopic (NICE), while the Japan NBI Expert Team (JNET) classification is used where endoscopy systems with optical magnification and the proper training is available. However, these classification systems have varying diagnostic accuracy and interobserver agreement. Previous prospective studies looking at CADx have utilized endocytoscopy and autofluorescence imaging (CAD-AFI) with positive results. However, the major limitation in these CADx studies is that these imaging systems are costly and are not readily available in most centres worldwide. Furthermore, most Clinicians performing colonoscopies have not been trained in these modalities of imaging and will have to rely completely on the CADx function to detect polyps if these imaging modalities are used, without being able to fall back on their experience and training should there be doubts about the accuracy of a CADx diagnosis in a real-world setting.

The Fujifilm 7000 System (Fujifilm Corp., Tokyo) has been in routine clinical use in all tertiary institutions in Singapore. The CAD EYE system was developed by Fujifilm Corp to aid Clinicians in colonoscopy with CADe and CADx functions. The basic functions and handling of the colonoscope, as well as the endoscopy processing unit, are similar to what is currently available in clinical practice, with the added CAD EYE software. The controller has been configured to allow the operator to activate and deactivate the CAD function depending on the need for it. These functions can be turned on and off using a button on the controller by the Clinician. The CADe and CADx functions operate when white light and blue laser imaging (BLI) are used, respectively. This provides a unique opportunity to externally validate the use of the CADx support tool by evaluating its diagnostic accuracy with final polyp histology as the gold standard, while also comparing its performance in a clinical setting against a Clinician using IEE (which is the conventional method of predicting polyp histology in colonoscopy).

The investigators plan to conduct a prospective, multi-centre clinical trial to validate the accuracy of CADx support for prediction of polyp histology in real-time colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have an indication for colonoscopy and who have at least one polyp detected during colonoscopy
2. 40 years of age and above
3. Consent obtained for the study

Exclusion Criteria:

1. Less than 39 years of age
2. Declined participation in study
3. Patients with no polyps detected during colonoscopy
4. Patients with inflammatory bowel disease
5. Patients with known unresected colorectal cancer

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients age 40 years and above and who have indications for colonoscopy will be eligible for the study. The patients who have been identified as eligible for the study will be counselled on the details, risks and benefits prior to the performance of colonoscopy. This counselling may take place in the outpatient or inpatient setting.
  Patients with one or more polyps detected during colonoscopy will be included in the study. The rest of the inclusion and exclusion criteria are as described.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of the CADx support tool compared to optical prediction of polyp histology by the Clinician in real-time colonoscopy in a clinical setting | 1 year
  Polyp histology used as gold standard

SECONDARY OUTCOMES:
To determine the diagnostic performance of CADx versus optical prediction of polyp histology by endoscopist in the subgroup analysis | 1 year
  Subgroups include bowel preparation, size of polyp and location

CONTACTS AND LOCATIONS:
Overall Officials: Dr James Li, Principal Investigator — Changi General Hospital, Singapore Health Services
Locations (1):
- Changi General Hospital, National University Hospital, Singapore General Hospital and Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Jemal A, Grey N, Ferlay J, Forman D. Global cancer transitions according to the Human Development Index (2008-2030): a population-based study. Lancet Oncol. 2012 Aug;13(8):790-801. doi: 10.1016/S1470-2045(12)70211-5. Epub 2012 Jun 1. PMID 22658655
- [Background] Araghi M, Soerjomataram I, Jenkins M, Brierley J, Morris E, Bray F, Arnold M. Global trends in colorectal cancer mortality: projections to the year 2035. Int J Cancer. 2019 Jun 15;144(12):2992-3000. doi: 10.1002/ijc.32055. Epub 2019 Jan 8. PMID 30536395
- [Background] Rex DK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Levin TR, Lieberman D, Robertson DJ. Colorectal Cancer Screening: Recommendations for Physicians and Patients from the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2017 Jul;112(7):1016-1030. doi: 10.1038/ajg.2017.174. Epub 2017 Jun 6. PMID 28555630
- [Background] Doubeni CA, Corley DA, Quinn VP, Jensen CD, Zauber AG, Goodman M, Johnson JR, Mehta SJ, Becerra TA, Zhao WK, Schottinger J, Doria-Rose VP, Levin TR, Weiss NS, Fletcher RH. Effectiveness of screening colonoscopy in reducing the risk of death from right and left colon cancer: a large community-based study. Gut. 2018 Feb;67(2):291-298. doi: 10.1136/gutjnl-2016-312712. Epub 2016 Oct 12. PMID 27733426
- [Background] Brenner H, Chang-Claude J, Jansen L, Knebel P, Stock C, Hoffmeister M. Reduced risk of colorectal cancer up to 10 years after screening, surveillance, or diagnostic colonoscopy. Gastroenterology. 2014 Mar;146(3):709-17. doi: 10.1053/j.gastro.2013.09.001. Epub 2013 Sep 5. PMID 24012982
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2017 Apr;49(4):378-397. doi: 10.1055/s-0043-103411. Epub 2017 Mar 7. PMID 28268235
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Vinsard DG, Mori Y, Misawa M, Kudo SE, Rastogi A, Bagci U, Rex DK, Wallace MB. Quality assurance of computer-aided detection and diagnosis in colonoscopy. Gastrointest Endosc. 2019 Jul;90(1):55-63. doi: 10.1016/j.gie.2019.03.019. Epub 2019 Mar 26. PMID 30926431
- [Background] Wang P, Liu X, Berzin TM, Glissen Brown JR, Liu P, Zhou C, Lei L, Li L, Guo Z, Lei S, Xiong F, Wang H, Song Y, Pan Y, Zhou G. Effect of a deep-learning computer-aided detection system on adenoma detection during colonoscopy (CADe-DB trial): a double-blind randomised study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):343-351. doi: 10.1016/S2468-1253(19)30411-X. Epub 2020 Jan 22. PMID 31981517
- [Background] Gong D, Wu L, Zhang J, Mu G, Shen L, Liu J, Wang Z, Zhou W, An P, Huang X, Jiang X, Li Y, Wan X, Hu S, Chen Y, Hu X, Xu Y, Zhu X, Li S, Yao L, He X, Chen D, Huang L, Wei X, Wang X, Yu H. Detection of colorectal adenomas with a real-time computer-aided system (ENDOANGEL): a randomised controlled study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):352-361. doi: 10.1016/S2468-1253(19)30413-3. Epub 2020 Jan 22. PMID 31981518
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Wang P, Berzin TM, Glissen Brown JR, Bharadwaj S, Becq A, Xiao X, Liu P, Li L, Song Y, Zhang D, Li Y, Xu G, Tu M, Liu X. Real-time automatic detection system increases colonoscopic polyp and adenoma detection rates: a prospective randomised controlled study. Gut. 2019 Oct;68(10):1813-1819. doi: 10.1136/gutjnl-2018-317500. Epub 2019 Feb 27. PMID 30814121
- [Background] Su JR, Li Z, Shao XJ, Ji CR, Ji R, Zhou RC, Li GC, Liu GQ, He YS, Zuo XL, Li YQ. Impact of a real-time automatic quality control system on colorectal polyp and adenoma detection: a prospective randomized controlled study (with videos). Gastrointest Endosc. 2020 Feb;91(2):415-424.e4. doi: 10.1016/j.gie.2019.08.026. Epub 2019 Aug 24. PMID 31454493
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Background] Repici A, Ciscato C, Correale L, Bisschops R, Bhandari P, Dekker E, Pech O, Radaelli F, Hassan C. Narrow-band Imaging International Colorectal Endoscopic Classification to predict polyp histology: REDEFINE study (with videos). Gastrointest Endosc. 2016 Sep;84(3):479-486.e3. doi: 10.1016/j.gie.2016.02.020. Epub 2016 Feb 27. PMID 26928372
- [Background] Komeda Y, Kashida H, Sakurai T, Asakuma Y, Tribonias G, Nagai T, Kono M, Minaga K, Takenaka M, Arizumi T, Hagiwara S, Matsui S, Watanabe T, Nishida N, Chikugo T, Chiba Y, Kudo M. Magnifying Narrow Band Imaging (NBI) for the Diagnosis of Localized Colorectal Lesions Using the Japan NBI Expert Team (JNET) Classification. Oncology. 2017;93 Suppl 1:49-54. doi: 10.1159/000481230. Epub 2017 Dec 20. PMID 29258091
- [Background] Kandel P, Wallace MB. Should We Resect and Discard Low Risk Diminutive Colon Polyps. Clin Endosc. 2019 May;52(3):239-246. doi: 10.5946/ce.2018.136. Epub 2019 Jan 21. PMID 30661337
- [Background] Neumann H, Neumann Sen H, Vieth M, Bisschops R, Thieringer F, Rahman KF, Gamstatter T, Tontini GE, Galle PR. Leaving colorectal polyps in place can be achieved with high accuracy using blue light imaging (BLI). United European Gastroenterol J. 2018 Aug;6(7):1099-1105. doi: 10.1177/2050640618769731. Epub 2018 May 17. PMID 30228899
- [Background] von Renteln D, Kaltenbach T, Rastogi A, Anderson JC, Rosch T, Soetikno R, Pohl H. Simplifying Resect and Discard Strategies for Real-Time Assessment of Diminutive Colorectal Polyps. Clin Gastroenterol Hepatol. 2018 May;16(5):706-714. doi: 10.1016/j.cgh.2017.11.036. Epub 2017 Nov 23. PMID 29174789
- [Background] Song EM, Park B, Ha CA, Hwang SW, Park SH, Yang DH, Ye BD, Myung SJ, Yang SK, Kim N, Byeon JS. Endoscopic diagnosis and treatment planning for colorectal polyps using a deep-learning model. Sci Rep. 2020 Jan 8;10(1):30. doi: 10.1038/s41598-019-56697-0. PMID 31913337
- [Background] Ang TL, Li JW, Wong YJ, Tan YJ, Fock KM, Tan MTK, Kwek ABE, Teo EK, Ang DS, Wang LM. A prospective randomized study of colonoscopy using blue laser imaging and white light imaging in detection and differentiation of colonic polyps. Endosc Int Open. 2019 Oct;7(10):E1207-E1213. doi: 10.1055/a-0982-3111. Epub 2019 Oct 1. PMID 31579701
- [Background] Mori Y, Kudo SE, Misawa M, Saito Y, Ikematsu H, Hotta K, Ohtsuka K, Urushibara F, Kataoka S, Ogawa Y, Maeda Y, Takeda K, Nakamura H, Ichimasa K, Kudo T, Hayashi T, Wakamura K, Ishida F, Inoue H, Itoh H, Oda M, Mori K. Real-Time Use of Artificial Intelligence in Identification of Diminutive Polyps During Colonoscopy: A Prospective Study. Ann Intern Med. 2018 Sep 18;169(6):357-366. doi: 10.7326/M18-0249. Epub 2018 Aug 14. PMID 30105375
- [Background] Horiuchi H, Tamai N, Kamba S, Inomata H, Ohya TR, Sumiyama K. Real-time computer-aided diagnosis of diminutive rectosigmoid polyps using an auto-fluorescence imaging system and novel color intensity analysis software. Scand J Gastroenterol. 2019 Jun;54(6):800-805. doi: 10.1080/00365521.2019.1627407. Epub 2019 Jun 14. PMID 31195905
- [Background] Byrne MF, Chapados N, Soudan F, Oertel C, Linares Perez M, Kelly R, Iqbal N, Chandelier F, Rex DK. Real-time differentiation of adenomatous and hyperplastic diminutive colorectal polyps during analysis of unaltered videos of standard colonoscopy using a deep learning model. Gut. 2019 Jan;68(1):94-100. doi: 10.1136/gutjnl-2017-314547. Epub 2017 Oct 24. PMID 29066576
- [Derived] Li JW, Wu CCH, Lee JWJ, Liang R, Soon GST, Wang LM, Koh XH, Koh CJ, Chew WD, Lin KW, Thian MY, Matthew R, Kim G, Khor CJL, Fock KM, Ang TL, So JBY; Artificial Intelligence in Gastrointestinal Endoscopy Singapore (AIGES) Study Group. Real-World Validation of a Computer-Aided Diagnosis System for Prediction of Polyp Histology in Colonoscopy: A Prospective Multicenter Study. Am J Gastroenterol. 2023 Aug 1;118(8):1353-1364. doi: 10.14309/ajg.0000000000002282. Epub 2023 Apr 11. PMID 37040553